CLINICAL TRIAL: NCT00238303
Title: Phase II Trial of Suberoylanilide Hydroxamic Acid (SAHA) in Patients With Recurrent Glioblastoma
Brief Title: Vorinostat in Treating Patients With Progressive or Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00646; NCI-2009-00646 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000445405; NCCTG-N047B; N047B (Other: North Central Cancer Treatment Group); N047B (Other: CTEP); U10CA025224 (NIH); NCT01647100 (obsolete NCT alias)
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2011-10

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Vorinostat; Surgical Procedures, Operative; Congresses as Topic

ARMS (2):
- Stratum 1 (not undergoing surgery) (Experimental): Patients receive oral vorinostat (SAHA) twice daily for 2 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Procedure: conventional surgery
- Stratum 2 (undergoing surgery) (Experimental): Beginning 3 days prior to surgery, patients receive oral SAHA once or twice daily for a total of 6 doses. Patients then undergo surgery to remove the tumor. Beginning within 1-4 weeks after surgery, patients receive oral SAHA twice daily for 2 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Procedure: conventional surgery

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Procedure: conventional surgery — Patients undergo surgery to remove tumor
  Other Names: surgery, conventional

SUMMARY:
This phase II trial is studying how well vorinostat works in treating patients with progressive or recurrent glioblastoma multiforme. Drugs used in chemotherapy, such as vorinostat, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving vorinostat before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving it after surgery may kill any remaining tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy of vorinostat (SAHA), in terms of 6-month progression-free survival, in patients with progressive or recurrent glioblastoma multiforme.

II. Determine the safety and toxicity of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics of this drug in these patients. II. Determine the biologic effect of this drug in target tissues, including primary tumor tissue, in these patients.

III. Correlate genetic alteration of tumors with response in patients treated with this drug.

OUTLINE: This is an open-label, multicenter study. Patients are stratified according to planned surgery (yes [stratum 1] vs no [stratum 2]) and number of prior chemotherapy regimens for progressive/recurrent disease (≤ 1 [stratum 1A] vs ≥ 2 [stratum 1B]).

STRATUM 1: Patients receive oral vorinostat (SAHA) twice daily for 2 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. (not undergoing surgery)

STRATUM 2: Beginning 3 days prior to surgery, patients receive oral SAHA once or twice daily for a total of 6 doses. Patients then undergo surgery to remove the tumor. Beginning within 1-4 weeks after surgery, patients receive oral SAHA twice daily for 2 weeks. (undergoing surgery)

Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed grade 4 astrocytoma (glioblastoma multiforme), including gliosarcoma, at primary diagnosis or recurrence

  * Progressive or recurrent disease
* Measurable or evaluable disease by MRI or CT scan
* Performance status - ECOG 0-2
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8 g/dL
* AST ≤ 3 times upper limit of normal (ULN)
* Bilirubin normal
* Creatinine ≤ 1.5 times ULN
* No myocardial infarction within the past 6 months
* No congestive heart failure
* No life-threatening ventricular arrhythmia requiring ongoing maintenance therapy
* No known HIV positivity
* Not immunocompromised except if related to the use of corticosteroids
* No known hypersensitivity to any of the components of the study drug
* No uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No other malignancy
* No other severe disease that would preclude study participation
* Prior adjuvant chemotherapy allowed
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* More than 2 weeks since prior small molecule cell cycle inhibitor
* Concurrent corticosteroids allowed as long as dose has been stable for ≥ 1 week
* At least 8 weeks since prior radiotherapy

  * Must have evidence of tumor progression by MRI or CT scan after radiotherapy
* More than 6 weeks since prior stereotactic radiosurgery or interstitial brachytherapy, unless 1 of the following criteria is met:

  * There is a separate lesion by MRI outside of the prior treatment field
  * There is evidence of recurrent disease by biopsy, MRI spectroscopy, or positron-emission tomography scan
* More than 2 weeks since prior valproic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2005-09; Primary Completion 2008-07 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 24 medical clinics in the United States between September 2005 to May 2008.
Groups:
- Stratum 1 (Not Undergoing Surgery): Patients not receiving pre-surgery SAHA with ≤1 prior chemotherapy regimens for progressive/recurrent disease. Patients receive oral vorinostat (SAHA) twice daily for 2 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  vorinostat : Given orally, 200 milligrams two times a day for 14 days followed by 7 days rest.
- Stratum 2 (Undergoing Surgery): Beginning 3 days prior to surgery, patients receive oral vorinostat (SAHA) once or twice daily for a total of 6 doses. Patients then undergo surgery to remove the tumor. Beginning within 1-4 weeks after surgery, patients receive oral SAHA twice daily for 2 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  vorinostat : Given orally, 200 milligrams two times a day for 14 days followed by 7 days rest.
  surgery : Patients undergo surgery to remove tumor
- Stratum 3 (Not Undergoing Surgery): Patients not receiving pre-surgery SAHA with ≥2 prior chemotherapy regimens for progressive/recurrent disease. Patients receive oral vorinostat (SAHA) twice daily for 2 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  vorinostat : Given orally, 200 milligrams two times a day for 14 days followed by 7 days rest.
Period: Overall Study
Arm/Group | Stratum 1 (Not Undergoing Surgery) | Stratum 2 (Undergoing Surgery) | Stratum 3 (Not Undergoing Surgery)
Started | 68 | 15 | 20
Completed | 53 | 13 | 11
Not Completed | 15 | 2 | 9
Not completed — Withdrawal by Subject | 11 | 1 | 2
Not completed — Death | 1 | 0 | 1
Not completed — Other Medical Problems | 2 | 0 | 2
Not completed — Poor tolerance of study treatment | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 (Not Undergoing Surgery) | Stratum 2 (Undergoing Surgery) | Stratum 3 (Not Undergoing Surgery) | Total
Number analyzed (Participants) | 68 | 15 | 20 | 103
Age, Continuous [Median (Full Range); unit: years] | 58 [26 to 78] | 49 [23 to 61] | 55.5 [25 to 78] | 56 [23 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 4 | 10 | 44
  Male | 38 | 11 | 10 | 59
Region of Enrollment [Number; unit: participants]
  United States | 68 | 15 | 20 | 103

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Successes (Patients Alive and Progression-free)
Description: Estimated using the Binomial point estimator (number of successes divided by the total number of evaluable patients) and the Binomial 95% confidence interval estimated by the exact method.
  Definition of progression:
  Bidimensionally measurable disease: >25% increase in product of perpendicular diameters of contrast enhancement or mass or appearance of new lesions.
  Evaluable disease (i.e., contrast enhancing mass on MRI and/or CT that is not bidimensionally measurable but clearly evaluable for response to therapy): unequivocal increase in size of contrast enhancement or increase in mass effect as agreed upon independently by primary physician and quality control physicians: appearance of new lesions.
Time Frame: At 6 months
Population: 68 Stratum 1 patients were enrolled. 2 stratum 1 patients did not receive treatment. Therefore, the remaining 66 patients were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Stratum 1 Patients That Started Treatment: Patients not receiving pre-surgery SAHA with ≤1 prior chemotherapy regimens for progressive/recurrent disease. Patients receive oral vorinostat (SAHA) twice daily for 2 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  vorinostat : Given orally, 200 milligrams two times a day for 14 days followed by 7 days rest.
Arm/Group | Stratum 1 Patients That Started Treatment | Stratum 2 (Undergoing Surgery) | Stratum 3 (Not Undergoing Surgery)
Number analyzed (Participants) | 66 | 15 | 20
percentage of participants | 15.2 [7.5 to 26.1] | 26.7 [7.8 to 55.1] | 10 [1.2 to 31.7]

2. Secondary Outcome: Survival
Description: Estimated using Kaplan-Meier survival curve.
Time Frame: From study registration to date of death due to any cause or last follow-up (up to 5 years)
Population: Stratum 1: 68 patients were enrolled. 2 patients did not receive treatment. Therefore, the remaining 66 patients were analyzed. The patient that survived 28 months was alive at last follow-up.
Measure: Median (Full Range); unit: months
Arm/Group | Stratum 1 (Not Undergoing Surgery) | Stratum 2 (Undergoing Surgery) | Stratum 3 (Not Undergoing Surgery)
Number analyzed (Participants) | 66 | 15 | 20
months | 5.7 [0.7 to 28] | 10.2 [2.8 to 41.6] | 2.2 [0.26 to 42.3]

3. Secondary Outcome: Confirmed Tumor Response
Description: A confirmed tumor response will be defined as an objective status of complete response (CR), partial response (PR), or regression (REGR) on two consecutive evaluations, which include neuroimaging, lasting during a period of at least 6 weeks. Confidence intervals for the true proportion will be calculated using the exact binomial method.
  Bidimensionally measurable disease:≥50% reduction in product of perpendicular diameters of contrast enhancement or mass with no new lesions with the patient being on stable or decreased steroid dose.
  Evaluable disease (i.e., contrast enhancing mass on MRI and/or CT that is not bidimensionally measurable but clearly evaluable for response to therapy): unequivocal reduction in size of contrast-enhancement or decrease in mass effect as agreed upon independently by primary physician and quality control physicians; no new lesions. Patient should be on stable or decreased steroid dose.
Time Frame: Assessed up to 5 years
Population: Stratum 1: 68 patients were enrolled. 2 patients did not receive treatment. Therefore, the remaining 66 patients were analyzed.
  Stratum 2: Since the patients underwent surgery, response is not applicable and hence 0 patients analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 1 (Not Undergoing Surgery) | Stratum 2 (Undergoing Surgery) | Stratum 3 (Not Undergoing Surgery)
Number analyzed (Participants) | 66 | 0 | 20
percentage of participants | 3.0 [0.4 to 10.5] |  | 0 [0 to 16.8]

4. Secondary Outcome: Time to Progression
Description: Estimated using Kaplan-Meier survival curve.
  Definition of progression:
  Bidimensionally measurable disease: >25% increase in product of perpendicular diameters of contrast enhancement or mass or appearance of new lesions.
  Evaluable disease (i.e., contrast enhancing mass on MRI and/or CT that is not bidimensionally measurable but clearly evaluable for response to therapy): unequivocal increase in size of contrast enhancement or increase in mass effect as agreed upon independently by primary physician and quality control physicians: appearance of new lesions.
Time Frame: From registration to disease progression (up to 5 years)
Population: Stratum 1: 68 patients were enrolled. 2 stratum 1 patients did not receive treatment. Therefore, the remaining 66 patients were analyzed. The patient that survived 28 months was progression-free at last follow-up.
Measure: Median (Full Range); unit: months
Arm/Group | Stratum 1 Patients That Started Treatment | Stratum 2 (Undergoing Surgery) | Stratum 3 (Not Undergoing Surgery)
Number analyzed (Participants) | 66 | 15 | 20
months | 1.9 [0.3 to 28] | 3.7 [1.4 to 41.6] | 1.4 [0.20 to 42.3]

ADVERSE EVENTS:
Groups:
- Stratum 1 (Not Undergoing Surgery); Stratum 3 (Not Undergoing Surgery): vorinostat : Given orally, 200 milligrams two times a day for 14 days followed by 7 days rest.
- Stratum 2 (Undergoing Surgery): surgery : Patients undergo surgery to remove tumor
Arm/Group | Stratum 1 (Not Undergoing Surgery) | Stratum 2 (Undergoing Surgery) | Stratum 3 (Not Undergoing Surgery)
Serious Adverse Events (participants affected / at risk) | 13/66 | 3/15 | 4/20
Other Adverse Events (participants affected / at risk) | 65/66 | 14/15 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 (Not Undergoing Surgery) (N=66) | Stratum 2 (Undergoing Surgery) (N=15) | Stratum 3 (Not Undergoing Surgery) (N=20)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 7 (7) | 0 (0) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 (Not Undergoing Surgery) (N=66) | Stratum 2 (Undergoing Surgery) (N=15) | Stratum 3 (Not Undergoing Surgery) (N=20)
Hemoglobin decreased (Blood and lymphatic system disorders) | 34 (156) | 10 (47) | 9 (57)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 12 (41) | 3 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (10) | 1 (11) | 2 (5)
Diarrhea (Gastrointestinal disorders) | 21 (63) | 7 (27) | 8 (12)
Dry mouth (Gastrointestinal disorders) | 2 (6) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Esophageal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 17 (52) | 8 (13) | 7 (15)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (14) | 4 (5) | 3 (4)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 3 (4) | 1 (2) | 0 (0)
Fatigue (General disorders) | 57 (192) | 11 (72) | 16 (46)
Fever (General disorders) | 2 (3) | 1 (3) | 0 (0)
Gait abnormal (General disorders) | 2 (2) | 0 (0) | 0 (0)
Localized edema (General disorders) | 2 (3) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gingival infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Penile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arterial injury - Extremity-lower (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (11) | 2 (3) | 3 (8)
Alkaline phosphatase increased (Investigations) | 7 (42) | 1 (1) | 2 (6)
Aspartate aminotransferase increased (Investigations) | 11 (19) | 2 (2) | 3 (8)
Blood bilirubin increased (Investigations) | 1 (1) | 3 (3) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (8)
Laboratory test abnormal (Investigations) | 1 (4) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 26 (109) | 9 (32) | 5 (31)
Lymphocyte count decreased (Investigations) | 5 (21) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 20 (87) | 6 (19) | 5 (16)
Platelet count decreased (Investigations) | 45 (198) | 12 (33) | 17 (55)
Serum cholesterol increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Weight gain (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 2 (2) | 1 (1) | 3 (9)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 18 (43) | 5 (22) | 10 (18)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 22 (37) | 1 (1) | 3 (37)
Dehydration (Metabolism and nutrition disorders) | 6 (10) | 2 (2) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 4 (6) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 4 (7) | 1 (1) | 1 (2)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (7)
Serum sodium increased (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0) | 3 (4)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (2)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Accessory nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 7 (9) | 0 (0) | 1 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 1 (4)
Depressed level of consciousness (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 5 (5) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 15 (51) | 3 (14) | 4 (6)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 12 (21) | 3 (3) | 2 (3)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0) | 1 (4)
Neurological disorder NOS (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 1 (34)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (11)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (6) | 0 (0)
Speech disorder (Nervous system disorders) | 7 (7) | 0 (0) | 1 (19)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 3 (4) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (4) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (4) | 1 (9) | 1 (1)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 2 (3) | 0 (0) | 1 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 2 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (7) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (21) | 1 (7) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less